CLINICAL TRIAL: NCT01705197
Title: A Double-blind, Stratified Randomization, Placebo Controlled, Parallel Group, Multicenter, Dose Escalation Study to Evaluate the Efficacy and Safety of Avanafil in Subjects With Moderate to Severe Erectile Dysfunction in Korea.
Brief Title: This Study is to Evaluate the Safety and Efficacy of Avanafil in the Treatment of Erectile Dysfunction.
Acronym: SPEED
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JW-AVA-302; 임상제도과-2221 (Other: KFDA)
Record Dates: First submitted 2012-09-26; First posted 2012-10-12 (Estimated); Last update posted 2017-03-10 (Actual); Status verified 2017-03

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Avanfil 100 or 200mg (Active Comparator): All subjects, who are judged to be suitable to the clinical trial after 4-week free run-in period was completed, should be administered with Avanafil 100mg(study group) or placebo 100mg(control group) for the first 4 weeks after randomization. When there are no moderate to severe adverse events at the 4 weeks evaluation after administration, and when it is decided by the researcher that the effect of Avanafil or placebo 100mg against erectile dysfunction is insufficient, a dosage increase to 200mg is executed. For subjects with a sufficient improvement effect on ED at 100mg, no dosage increase is allowed, and the previous 100mg administration should be maintained until the termination of the study.
  Interventions: Drug: Avanafil 100 or 200mg
- Placebo 100mg or 200mg (Placebo Comparator): When there are no moderate to severe adverse events at the 4 weeks evaluation after administration, and when it is decided by the researcher that the effect of Avanafil or placebo 100mg against erectile dysfunction is insufficient, a dosage increase to 200mg is executed.
  Interventions: Drug: Avanafil 100 or 200mg

INTERVENTIONS:
Drug: Avanafil 100 or 200mg — This study is designed as a double-blind, stratified randomized, placebo controlled, parallel group, multicenter, dose escalation study. For subjects with moderate to severe ED who have voluntarily signed the consent form, conduct screening and undertake the 4 weeks Free run-in period. For those who satisfy the study criteria during the review of subject's diaries composed during the free run-in period and the evaluation of inclusion/exclusion criteria at a future visit, drugs for each group are provided after randomized to Avanafil 100mg or placebo 100mg at a ratio of 2:1. At this time, subjects are random stratified to each group depending on their diabetes status.
  Other Names: Zepeed 100mg or 200mg

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of Avanafil in the treatment of erectile dysfunction with moderate to severe in subjects. And, this is to additionally confirm the efficacy and safety after initiating treatment with Avanafil 100mg and later increasing to 200mg, compared with continuing treatment with Avanafile 100mg, in subjects.

DETAILED DESCRIPTION:
All subjects, who are judged to be suitable to the clinical trial after 4-week free run-in period was completed, should be administered with Avanafil 100mg(study group) or placebo 100mg(control group) for the first 4 weeks after randomization. When there are no moderate to severe adverse events at the 4 weeks evaluation after administration, and when it is decided by the researcher that the effect of Avanafil or placebo 100mg against erectile dysfunction is insufficient, a dosage increase to 200mg is executed. For subjects with a sufficient improvement effect on ED at 100mg, no dosage increase is allowed, and the previous 100mg administration should be maintained until the termination of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male patients over 20 years old with a history of erectile dysfunction for at least 6 months prior to participation in the study
2. Patients in a stable relationship with 1 female partner
3. Patients whose sex partner is not in pregnancy or lactating, and is taking proper contraceptive
4. Patients who have voluntarily decided to participate in this clinical trial, and signed the informed consent form
5. Patients whose failure rate for sexual intercourse is more than 50% after attempts of sexual intercourse on more than 3 different days (once/day) at least during the 4-week Free run-in period
6. Patients whose EF domain score is less than 18 points (moderate to severe erectile dysfunction) in the IIEF questionnaire after the 4-week Free run-in period

Exclusion Criteria:

1. Patients who have a spinal injury or have had a radical prostatectomy
2. Patients with anatomical malformations of the penis (example: angulation, fibrosis of corpus cavernosum, peyronies disease, etc.)
3. Patients who had surgery in the pelvic cavity within 6 months prior to participation in the study
4. Patients with neurogenic or endocrine (example: hyperprolactinemia, low testosterone, etc.) ED

   * Hyperprolactinemia: Serum prolactin ≥ 3 X ULN
   * Low testosterone: Total testosterone is less than the normal lower limit(testosterone is susceptible to daily changes, so enrollment is permitted after retesting before 11 am, only limited to once, when the number is 20% less than the normal lower limit.)
5. Patients with a major refractory psychiatric disorder (including major depression or schizophrenia) or significant neurological abnormalities (neurovascular disease)
6. Patients with alcohol addiction or persistent abuse of drugs of dependence
7. Patients with hepatic dysfunction or renal dysfunction as per the following:

   * Hepatic dysfunction: AST, ALT ≥ 3 X ULN
   * Renal dysfunction: Serum creatinine > 2.0mg/dL
8. Diabetic patients whose HbA1c exceeds 12%
9. Patients with proliferative diabetic retinopathy
10. Patients who have had a stroke, TIA(Transient ischemic attack), MI(Myocardial Infarction) or fatal arrhythmia, or severe heart failure, unstable angina or who underwent coronary artery bypass grafting (CABG) within the last 6 months prior to participation in the study
11. Patients with hypotension (resting SBP/DBP in the sitting position is less than 90/50mmHg) or unregulated hypertension (resting SBP/DBP in the sitting position exceeds 170/100mmHg)
12. Patients with hematopathy, which can be a predisposition to priapism (sickle-cell disease, multiple myeloma, leukemia)
13. Patients with a known genetically degenerative retinopathy, including retinitis pigmentosa
14. Patients who have had experience with avanafil, viagra, cialis, levitra, yaila, zydena, mvix or other ED treatment within 2 weeks from participation in the study
15. Patients administered with the following medications:

    * Nitrate/Nitric oxide (NO) donors (example: nitroglycerin, isosorbide mononitrate, amyl nitrate/nitrite, sodium nitroprusside)
    * Androgens (example: testosterone), anti-androgen, trazodone
    * Anticoagulant (antiplatelet agents excluded)
    * Agents that significantly affect the CYP450 3A4 intermediary metabolism, such as erythromycin, intraconazol, ketoconazol, cimetidine, ritonavir, saquinavir, amprenavir, indinavir, and nelfinavir, etc.
16. Patients who have had a history of hypersensitivity to other PDE-5 inhibitors or who have not responded to them
17. Patients with primary hyposexuality
18. Patients who have taken other investigational products within 4 weeks before the study
19. For other reasons besides the aforementioned cases, patient whose participation is deemed inappropriate due to clinically significant findings according to the medical decision of the principal investigator or the study personnel

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2012-02; Primary Completion 2013-04 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Compare with the changes in IIEF(The International Index of Erectile Function)Erectile Function domain score between the study group and control group. | 12 weeks
  When changes in IIEF EF domain score of the study group (Avanafil-administered group) and control group (placebo-administered group) are compared to the baseline after 12 weeks post medication, it is to evaluate the superiority of the study group.

SECONDARY OUTCOMES:
Compare with the MSHQ, SEP Q2, SEP Q3 and GEAQ. | 12 weeks
  1. When a dose is increased to 200mg because the effect is insufficient after 4 weeks of medication with Avanafil 100mg, it is to evaluate the effect of a dosage increase in IIEF EF domain, SEP Q2 and Q3.
  2. It is to evaluate changes in SEP (Q2, Q3, Q4 and Q5), other domains of IIEF (such as OF, SD, IS and OS domain), IIEF Q3, IIEF Q4, MSHQ, rate of subjects who score 26 and over in EF domain, GEAQ of the study group and control group compared to the baseline after 12 weeks post medication.
  3. Change in total score of IIEF EF domain, SEP Q2 and Q3; Comparison between the result from the 12th week and the result from the baseline and the 4th week.
  [Glossary] MSHQ: Male Sexual Health Questionnaire SEP: Sexual Encounter Profile SEP Q2: Intercourse success rates on the Sexual Encounter Profile SEP Q3: Erectile success rates on the Sexual Encounter Profile GEAQ:Global Assessment Question

OTHER OUTCOMES:
We will be confirming the safety after initiating treatment with Avanafil 100mg and later increasing to 200mg, compared with continuing treatment with Avanafil 100mg. | 12weeks
  1. Comparative evaluate the variables of the study group and control group after medication: physical exam, vital sign(BP, pulse), ECG(Electrocardiogram, ECG=EKG), Laboratory tests, Adverse events
  2. We will check or confirm adverse events related to rates of adverse drug reactions and the disappearance time of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Se Woong, Doctor, Principal Investigator — Catholic hospital in Korea
Locations (1):
- Catholic Univ. Seoul St. Mary's Hospital, Seoul, South Korea